CLINICAL TRIAL: NCT01494467
Title: A Phase 3 Randomized, Double Blind, 12 Week Vehicle Controlled, Parallel Group Study Assessing the Efficacy and Safety of CD5024 1 % Cream Versus Vehicle Cream in Subjects With Papulopustular Rosacea, Followed by a 40 Week Investigator Blinded Extension Comparing the Long Term Safety of CD5024 1% Cream Versus Azelaic Acid 15 % Gel.
Brief Title: Phase 3 Papulopustular Rosacea Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18171
Record Dates: First submitted 2011-12-14; First posted 2011-12-19 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2015-01

CONDITIONS: Papulopustular Rosacea
Keywords: PPR
MeSH Terms: conditions — Rosacea | interventions — azelaic acid; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CD5024 (Experimental): CD5024 1% Cream
  Interventions: Drug: CD5024
- CD5024 Vehicle (Placebo Comparator): CD5024 Vehicle Cream
  Interventions: Drug: Azelaic acid 15% Gel

INTERVENTIONS:
Drug: CD5024 — CD5024 1% Cream, once daily
  Arms: CD5024
Drug: Azelaic acid 15% Gel — Topical Gel applied twice daily
  Arms: CD5024 Vehicle

SUMMARY:
The purpose of this study is to demonstrate that CD5024 1% cream is more effective than its vehicle when applied once daily, at bed time, during a 12 week period in subjects with Papulopustular Rosacea (PPR) and continues to be safe up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has papulopustular rosacea with an Investigator Global Assessment (IGA) score rated 3 (moderate) or 4 (severe),
2. The subject has at least 15 but not more than 70 inflammatory lesions (papules and pustules) on the face.

Exclusion Criteria:

1. The subject has particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) or other facial dermatoses that may be confounded with papulopustular rosacea, such as peri oral dermatitis, facial keratosis pilaris, seborrheic dermatitis, and acne,
2. The subject has rosacea with more than two nodules on the face.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2011-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, M.D., Study Director — Galderma R&D, LLC
Locations (50):
- United States (40):
  - Total Skin and Beauty, Birmingham, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Dermatology Specialists, Inc, Oceanside, California
  - Integrated Research Group, Inc, Riverside, California
  - Therapeutics Clinical Research, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - ATS Clinical Research, Santa Monica, California
  - Redwood Dermatology Research, Santa Rosa, California
  - FXM Research Corp Miami, Miami, Florida
  - Leavitt Medical Associates of Florida dba Ameriderm Research, Ormond Beach, Florida
  - Atlanta Dermatology, Vein & Research Center, LLC, Alpharetta, Georgia
  - Emory University, Atlanta, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Northwestern University, Chicago, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dermatology Specialists Research, Louisville, Kentucky
  - Northeast Dermatology Associates, Beverly, Massachusetts
  - David Fivenson, MD, PLC, Ann Arbor, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Dermatology Clinical Trials Unit, St Louis, Missouri
  - Psoriasis Treatment Center of NJ, West Windsor, New Jersey
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - DermResearch Center of New York, Inc, Stony Brook, New York
  - High Point, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Dermatology and Skin Surgery Center, Exton, Pennsylvania
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Paddington Research, Philadelphia, Pennsylvania
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - The Skin Wellness Center, Knoxville, Tennessee
  - Dermatology Reserach Associates, Nashville, Tennessee
  - Arlington Research Center, Inc, Arlington, Texas
  - Stephen Miller MD, San Antonio, Texas
  - San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
- Canada (10):
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - Ultranova Skincare, Barrie, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - The Guenther Dermatology Research Center, London, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - North Bay Dermatology Centre, Inc, North Bay, Ontario
  - The Centre for Dermatology & Cosmetic Surgery, Richmond Hill, Ontario
  - XLR8 Medical Research, Inc, Windsor, Ontario
  - International Dermatology Research, Inc, Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec Metropolitan, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- CD5024 1% Cream: Part A & B: CD5024 1% Cream, once daily application
- CD5024 Vehicle Cream/Azelaic Acid 15% Gel: Part A: CD5024 Vehicle Cream, once daily application
  Part B: Azelaic acid 15% Gel, twice daily application
Period: Part A Vehicle Control (12 Weeks)
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream/Azelaic Acid 15% Gel
Started | 459 | 229
Completed | 429 | 208
Not Completed | 30 | 21
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 6 | 4
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Protocol Violation | 4 | 0
Not completed — Lost to Follow-up | 8 | 8
Not completed — Other | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Period: Part B Long Term Active Control 40 Weeks
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream/Azelaic Acid 15% Gel
Started | 428 (429 completed Part A. Subsequently, one subject discontinued so only 428 entered Part B) | 208
Completed | 353 | 159
Not Completed | 75 | 49
Not completed — Pregnancy | 2 | 0
Not completed — Lack of Efficacy | 1 | 3
Not completed — Adverse Event | 3 | 5
Not completed — Withdrawal by Subject | 32 | 24
Not completed — Protocol Violation | 3 | 5
Not completed — Lost to Follow-up | 26 | 10
Not completed — Other (noted in eCRF) | 8 | 2
Period: Part C Safety Follow up (4 Weeks)
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream/Azelaic Acid 15% Gel
Started | 353 | 159
Completed | 353 | 159
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- CD5024 1% Cream: Part A: CD5024 1% Cream, once daily application for 12 weeks
  Part B: CD5024 1% Cream, once daily application for 40 weeks
- CD5024 Vehicle Cream/Azelaic Acid 15% Gel: Part A: CD5024 Vehicle Cream, once daily application for 12 weeks
  Part B: Azelaic acid 15% Gel, twice daily application for 40 weeks
- Total: Total of all reporting groups
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream/Azelaic Acid 15% Gel | Total
Number analyzed (Participants) | 459 | 229 | 688
Age, Continuous [Mean (Standard Deviation); unit: Year] | 50.5 (12.35) | 49.5 (12.16) | 50.2 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 145 | 459
  Male | 145 | 84 | 229
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 31 | 87
  Not Hispanic or Latino | 403 | 198 | 601
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 438 | 218 | 656
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Skin Photo Type [Number; unit: Participants] — DEFINITION OF SKIN PHOTOTYPE (T.B. Fitzpatrick):
  I: Always burns easily ; never tans II: Always burns easily ; tans minimally and with difficulty III: Burns minimally ; tans gradually and uniformly (light Brown) IV: Burns minimally ; always tans well (moderate brown) V: Rarely burns ; tans profusely (dark brown)) VI:Never burns ; deeply pigmented (black), tans profusely
  Participants
    I | 48 | 22 | 70
    II | 211 | 96 | 307
    III | 139 | 71 | 210
    IV | 50 | 31 | 81
    V | 11 | 7 | 18
    VI | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: Percentage of subjects who achieve "Clear" (Score 0) or "Almost Clear" (Score 1) at Week 12 (ITT-LOCF) based on the Investigator Global Assessment (IGA) Score.
  Evaluation of papulopustular rosacea will be performed by the investigator based on the following 5 point scale:
  Clear = 0 (No inflammatory lesions present, no erythema); Almost Clear = 1 (Very few small papules/pustules, very mild erythema present); Mild = 2 (Few small papules/pustules, mild erythema); Moderate = 3 (Several small or large papules/pustules, moderate erythema); Severe = 4 (Numerous small and/or large papules/pustules, severe erythema)
Time Frame: Week 12
Population: LOCF, ITT
Measure: Number; unit: Percentage of participants
Groups:
- CD5024 1% Cream: CD5024 1% Cream, once daily application for 12 weeks
- CD5024 Vehicle Cream: CD5024 Vehicle Cream, once daily application for 12 weeks
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream
Number analyzed (Participants) | 459 | 229
Percentage of participants | 40.1 | 18.8
Statistical Analysis 1: Comparison: CD5024 1% Cream vs CD5024 Vehicle Cream; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Primary Outcome: Absolute Change in Inflammatory Lesion Count
Description: Inflammatory lesion counts were conducted at each visit by the Investigator or study coordinator. Papules and pustules were counted separately on each of the five facial regions (forehead, chin, nose, right cheek, left cheek).
Time Frame: Baseline to Week 12
Population: LOCF, ITT
Measure: Mean (Standard Deviation); unit: Lesion count change
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream
Number analyzed (Participants) | 459 | 229
Lesion count change | -22.2 (14.87) | -13.4 (14.48)
Statistical Analysis 1: Comparison: CD5024 1% Cream vs CD5024 Vehicle Cream; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -8.22, 95% CI 2-sided [-10.18 to -6.25]

3. Secondary Outcome: Percent Change in Inflammatory Lesion Count From Baseline to Week 12 (ITT-LOCF)
Description: as for outcome 2
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: Percentage of change in lesion counts
Arm/Group | CD5024 1% Cream | CD5024 Vehicle Cream
Number analyzed (Participants) | 459 | 229
Percentage of change in lesion counts | -65.7 (33.18) | -43.4 (38.42)
Statistical Analysis 1: Comparison: CD5024 1% Cream vs CD5024 Vehicle Cream; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Time of signed informed consent to study end (~ 58 wks). Treatment emergent adverse events - occurred on date of 1st use of medication or after, except those reported from Day 1 lab data as blood sample was to be drawn before the time of 1st dose.
Description: Number of participants at risk based on actual number of participants who received each intervention as randomized or due to dispensing errors (3 subjects).
Groups:
- CD5024 1% Cream - Part A: Part A: CD5024 1% Cream, once daily application for 12 weeks
- CD5024 Vehicle Cream - Part A: Part A: CD5024 Vehicle Cream, once daily application for 12 weeks
- CD5024 1% Cream - Part B: Part B CD5024 1% Cream, once daily application for 40 weeks
- Azelaic Acid 15% Gel - Part B: Part B: Subjects in the CD5024 Vehicle Cream arm applied Azelaic Acid 15% Gel twice daily for 40 weeks
- CD5024 1% Cream - Part C; CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Part C: Part C: 4 week safety follow up. No drug applications
- CD5024 1% Cream - Overall; CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Overall: Overall number of subjects with adverse events for the entire duration of study
Arm/Group | CD5024 1% Cream - Part A | CD5024 Vehicle Cream - Part A | CD5024 1% Cream - Part B | Azelaic Acid 15% Gel - Part B | CD5024 1% Cream - Part C | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Part C | CD5024 1% Cream - Overall | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Overall
Serious Adverse Events (participants affected / at risk) | 7/458 | 4/230 | 13/428 | 4/208 | 0/353 | 1/159 | 18/460 | 9/231
Other Adverse Events (participants affected / at risk) | 33/458 | 26/230 | 102/428 | 47/208 | 4/353 | 3/159 | 125/460 | 64/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD5024 1% Cream - Part A (N=458) | CD5024 Vehicle Cream - Part A (N=230) | CD5024 1% Cream - Part B (N=428) | Azelaic Acid 15% Gel - Part B (N=208) | CD5024 1% Cream - Part C (N=353) | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Part C (N=159) | CD5024 1% Cream - Overall (N=460) | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Overall (N=231)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD5024 1% Cream - Part A (N=458) | CD5024 Vehicle Cream - Part A (N=230) | CD5024 1% Cream - Part B (N=428) | Azelaic Acid 15% Gel - Part B (N=208) | CD5024 1% Cream - Part C (N=353) | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Part C (N=159) | CD5024 1% Cream - Overall (N=460) | CD5024 Vehicle Cream/Azelaic Acid 15% Gel - Overall (N=231)
Nasopharyngitis (Infections and infestations) | 10 | 6 | 43 | 18 | 1 | 1 | 52 | 23
Upper respiratory tract infection (Infections and infestations) | 12 | 8 | 40 | 17 | 1 | 2 | 48 | 23
Sinusitis (Infections and infestations) | 9 | 6 | 20 | 7 | 2 | 0 | 30 | 13
Skin irritation (Skin and subcutaneous tissue disorders) | 3 | 7 | 4 | 8 | 0 | 0 | 6 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty (60) days prior to submission for publication, presentation or use, the Institution and the Investigator shall submit in writing to the Contract Research Organization and Sponsor for review and comment any proposed oral or written publication, which period may be extended for an additional thirty (30) days if requested in writing by Contract Research Organization and Sponsor.